CLINICAL TRIAL: NCT02555904
Title: Do VoIce Changes Predict Heart Failure
Brief Title: VoIce Changes and Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Marc Semigran, Physician investigator, Massachusetts General Hospital
Other Study IDs: 2015P000986
Record Dates: First submitted 2015-09-18; First posted 2015-09-22 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Heart Failure; Voice; Congestion; Pitch
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart failure syndrome & pulmonary congestion: Patients who are admitted for inpatient management with acute heart failure syndrome with pulmonary congestion who require intravenous diuretics are potential candidates for the study and shall be screened for suitability based on the inclusion and exclusion criteria.

SUMMARY:
This is an observational, single center study to evaluate if acoustic and accelerometer-based measures of voice and speech have sufficient precision to detect a change in lung fluid status for patients with confirmed acute heart failure syndrome with pulmonary congestion. The study shall be conducted in concordance with the United States FDA regulations for a non-significant risk study. Patients admitted for acute heart failure syndrome with pulmonary congestion with an expected stay greater than 3 to 4 days, who are willing and able to sign an informed consent, and who meet all inclusion/exclusion criteria, as identified by the clinical investigator, will be enrolled in the study. Results of this study will evaluate the sensitivity of voice and speech measures in detecting changes in lung fluid status in a symptomatic population. Up to 12 subjects will be enrolled to comparatively evaluate the voice outcome measures in this pilot study.

DETAILED DESCRIPTION:
There are two specific aims for this first phase of the project:

1. Collect short-term acoustic and accelerometric data on groups of patients with volume overload before and after successful diuresis of amounts of fluid that are large enough to permit robust statistical testing of derived measures.
2. Determine whether direct measures (based on previously-developed approaches for acoustic and ACC-based monitoring of vocal function can differentiate between hypervolemic and optivolemic patterns.

2.2 Justification for Clinical Study The study will evaluate if acoustic and accelerometric measures of voice and speech production have the sensitivity to detect a clinically significant change in lung fluid status for patients with confirmed acute heart failure syndrome with pulmonary congestion. Changes in lung fluid in acute heart failure syndrome are difficult to diagnose and evaluate. A blinded observational methodology was chosen as the most appropriate study design to understand changes in lung fluid values in patients with acute heart failure syndrome with pulmonary congestion. The primary endpoint is significant correlation of changes in voice and speech characteristics with change in total body water as measured by change in weight during the hospital admission.

2.3 Measurement Precision Exploratory endpoints will be to determine the distributions of lung fluid values for patients with confirmed acute heart failure syndrome and to determine if acoustic and accelerometer-based measurements have sufficient sensitivity to detect changes in lung fluid status in a symptomatic hospitalized population. The establishment of the underlying etiology of the heart failure will help determine how it may contribute to symptomology and changes in acoustic and accelerometric measures of voice and speech production. The types of analyses that can be performed on the airborne acoustic (microphone) signal are somewhat limited by the levels of background noise in the recording environment, particularly with respect to some of the acoustic measures related to voice quality. For this reason it is proposed that recordings of voice/speech production for this pilot study be obtained simultaneously with both a microphone and a neck-placed miniature accelerometer (ACC). The ACC is relatively immune to environmental noise, and we have been able to extract some voice quality-related measures from the ACC signal. The ACC is easily placed on the anterior neck just above the clavicular notch using double-sided medical grade adhesive tape (see Figure 1). The recording protocol will be comprised of: 1) sustained vowels, 2) standard sentences and a reading passage, and 3) 30 seconds of spontaneous speech. Recordings will be made before, during, and after an acute episode of Congestive Heart Failure (CHF). Each recording session should take less than 10 minutes.

3 STUDY PROTOCOL 3.1 Study Design and Objective - see above

3.2 Study Duration Enrollment in the trial is expected to take approximately 4 months including enrollment.

3.2.1 Enrollment Procedure and Follow-up Procedure Patients will be screened and enrolled prior to admission required for their medical management. Subjects enrolled in the study will have their baseline voice recordings made within 24 hours of admission. Following their index measurement, all subjects will have their recording performed daily within the first 96 hours and on discharge and/re reaching presumed dry weight. At the discretion of the investigator, voice recordings may be obtained more frequently but no more than once per day of the hospital admission up to a maximum of ten (10) days.

Inclusion and Exclusion Criteria: see below

4.0 OutComes - See below for primary and secondary endpoints

5 Statistical Methods 5.1 Introduction This is an observational study. Subjects are enrolled in the study throughout their inpatient stay up to maximum of 10 days. The objective of the statistical analysis is to determine via Pearson correlation if voice and speech measures have sufficient precision to detect clinically significant changes in overall volume status for those experiencing acute heart failure syndromes.

5.2 Confirmation of a reduction in body fluid volume In order to confirm that a clinically significant reduction in overall volume status has occurred during the voice recording period, a cardiologist will review all relevant medical records pertaining to the patient and independently determine if the admission resulted in reduction in volume overload. They will have access to source medical records and any additional information that becomes available after the evaluation in the hospital environment. This information will include the following: reading of the chest roentgenograms obtained in the emergency department or inpatient stay by a radiologist, medical history obtained from a medical chart that was not available to the emergency department physicians at the time of presentation, the results of subsequent tests, such as echocardiography, radionuclide angiography,or left ventriculography, performed at the time of cardiac catheterization, and the hospital course for patients admitted to the hospital.

6 Statistical Analysis 6.1. Data Analyses

Digital signal processing approaches will be to extract the following measures from the acoustic and ACC signals:

A. Sustained vowels: measures related to voice quality including perturbation (jitter and shimmer) and signal-to-noise levels (harmonics-to-noise, spectral, and cepstral measures), and the frequency locations of subglottal resonances.

B. Connected speech (sentences, reading, and spontaneous speech): measures related to sound segment, suprasegmental, and utterance length parameters including pitch (fundamental frequency), loudness (relative sound pressure level), and articulation/timing (sound segment durations, vocalic formant transitions, pauses).

7 Study Visits 7.1 Pre-Enrollment Evaluations and Parameters

Pre-enrollment procedures and protocols for all subjects will follow the standard hospital practice but should, at a minimum, include the following:

* Subject demographics
* History and physical exam, including weight
* Medical history
* Dyspnea as quantified by the VAS instrument
* Blood NT-proBNP level

7.2 During Enrollment

* Voice assessment
* Weight and other vital signs
* Dyspnea visual analog scale (DVAS)
* Global assessment of symptoms (GVAS)
* N-terminal pro-brain natriuretic peptide NTproBNP

7.3 At Discharge (or when deemed to be at dry weight) assessment (max 10 days post admission)

* Voice assessment
* Weight and other vital signs
* Dyspnea visual analog scale (DVAS)
* Global assessment of symptoms (GVAS)
* (NTproBNP)

ELIGIBILITY:
Inclusion Criteria:

* • > 18 years

  * Prior diagnosis of heart failure with daily use of loop diuretic
  * Must be identified within 48 hrs of admission
  * Diagnosis of acute Congestive Heart Failure (CHF) as defined by at least one symptom or one clinical sign
  * Believed to be > 10 lbs above target weight
  * Anticipated need for iv loop diuretic for at least 48 hrs

Exclusion Criteria:

* Inability to perform VA

  * Respiratory infection
  * Significant pulmonary disease requiring the use of inhaler bronchodilators or steroids
  * Anticipate need for vasoactive agent or ultrafiltration
  * Systolic BP < 90 mmHg
  * Serum Cr > 3 on admission or requirement for dialysis
  * Hemodynamically significant arrhythmias
  * Acute Coronary Syndrome (ACS) within 4 weeks
  * Hypertrophic Obstructive Cardiomyopathy (HOCM)
  * Severe stenotic valve disease
  * Complex congenital heart disease
  * Sepsis
  * Active smoking within 1 year
  * O2 saturation less than 92% on room air
  * History of diagnosed vocal cord pathology / dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute heart failure syndromes admitted for inpatient management meeting inclusion and exclusion criteria will be asked to consent for the study.
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Relationship between change in pitch and change in total body water | 10 days
  correlation of change in fundamental frequency with change in weight

SECONDARY OUTCOMES:
relationship between change in pitch and change in NTproBNP | 10 days
  change in fundamental frequency correlates with change in plasma NTproBNP levels
correlation in change in pitch with change in dyspnea visual analog scale (DVAS) | 10 days
  correlation in change in fundamental frequency with change in DVAS

CONTACTS AND LOCATIONS:
Overall Officials: Marc Semigran, MD, Principal Investigator — Massachusetts General Hospital